CLINICAL TRIAL: NCT05467956
Title: The Incidence of AKI in Critically-ill COVID -19 Patients, A Single Centre Retrospective Study From March 2020 Till September 2021.
Brief Title: Incidence of Acute Kidney Injury in Covid-19
Acronym: COVIDAKI
Status: Completed | Type: Observational
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Sponsor
Other Study IDs: MREC#2602
Record Dates: First submitted 2022-07-20; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Acute Kidney Injury; COVID-19; Critically Ill
Keywords: Acute Kidney Injury; COVID-19; renal replacement therapy; hyperglycemia; incidence; risk factors
MeSH Terms: conditions — Acute Kidney Injury; COVID-19; Critical Illness; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Covid-19 — Covid-19 disease

SUMMARY:
Acute kidney injury (AKI) in Covid-19 patients is a topic that receives little attention in the literature, although being important in clinical practice in the ICU, particularly in Oman. Our objective was to determine the incidence of AKI, risk factors, and the requirement of renal replacement treatment.

Methods: All adult patients hospitalized at Sultan Qaboos University Hospital in the critical care unit (ICU) between March 2020 and September 2021 with laboratory-confirmed Covid-19 had their medical records retrospectively reviewed. All patient characteristics, their course of events, and the treatment received in ICU were noted.

The incidence of AKI, its association with the glycemic index, and other possible risk factors will be studied. Those requiring renal replacement therapy will be studied in terms of its predictors and outcomes.

DETAILED DESCRIPTION:
Throughout the world, Coronavirus disease 2019 (COVID-19) is spreading as a pandemic disease. Asymptomatic viral carriers to critically ill patients are found to be affected by Covid-19, which has diverse clinical manifestations. There have been an increase in hospitalizations, respiratory failure, and intensive care unit (ICU) admissions due to this disease.

It has been reported that acute kidney injury (AKI) is a common complication of COVID-19 that is associated with a higher mortality rate. It has been reported that AKI in patients with COVID-19 infection ranges from 6.5% to 46% [3], with the highest rates among critically ill patients (23%-81%]. Different definitions of AKI and different populations have resulted in different incidences of AKI.

Several factors have been suggested as contributing to the development of AKI in patients with COVID-19: immunologic injury associated with inflammatory response, direct cytotoxicity over endothelial and tubulo-epithelial cells and podocytes, microthrombi and thrombotic microangiopathy, or cardiorenal syndrome due to right ventricular failure may be present.

There are limited studies in the middle east, especially in Oman, investigating the incidence of AKI in critically ill COVID-19 patients. The aim of this study is to investigate the incidence of AKI, the possible predictive factors for its occurrence in critically ill COVID-19 patients, and the requirement of renal replacement therapy (RRT).

This is a retrospective cohort study carried out in the University hospital in Oman, Sultan Qaboos University Hospital (SQUH), between March 2020 to September 2021. All adult patients admitted to ICU with laboratory-confirmed SARS-CoV-2 infection, documented by real-time RT-PCR on nasopharyngeal swabs, or lower respiratory tract aspirates were included.

Patients with the pre-existing renal disease with eGFR< 30 or on dialysis and insufficient clinical documentation available for review were excluded. Data was obtained from SQUH "Track Care" hospital information system.

Sample size The sample size was estimated based on the expected incidence proportion of AKI among COVD-19 patients. A recently published systematic review has reported a pooled incidence proportion of 19.45% (95% CI: 14.63 - 24.77)[5]. Therefore, the estimated sample size is based on an expected incidence proportion of 20%, a margin of error of 5%, and a confidence level of 95%. The estimated sample size was 250.

Definition of acute kidney injury Kidney Disease Improving Global Outcomes (KDIGO) criteria were used for AKI diagnosis and stratification: stage 1 - increase in serum creatinine from 0.3 mg/dL in 48 hours or increase from 1.5 to 1.9 value of baseline serum creatinine within 7 days; stage 2 - 2 to 2.9-fold increase in serum creatinine within 7 days or urine output below 0.5 mL/kg/h for more than 12 hours; and stage 3 - 3-fold increase in serum creatinine in 7 days or creatinine higher than 4 mg/dL or the initiation of renal replacement therapy through hemodialysis or urine output below 0.3 mL/kg/h for 24 hours or more, or anuria for 12 hours or more. On admission to the ICU, the level of creatinine was measured as a baseline.

Data collection:

To describe the population's characteristics, The following data were used: age, sex, BMI (kg/m2), hypertension (HTN), diabetes mellitus (DM), lung illness (asthma, COPD), cardiovascular disease, chronic kidney disease, onset, length of ICU stay, ventilator days, shock, nephrotoxic agents, the patient medications for DM and details of renal replacement therapy.

Laboratory tests were collected upon admission to the ICU, including PF ratio, full blood count, inflammatory markers (C-reactive protein, IL-6, and ferritin), blood sugar level, D-dimer, and Electrolytes.

All data will be entered into an Excel file and kept under lock. The patient's identity was coded and the complete data file was shared with the statistician.

ELIGIBILITY:
Inclusion Criteria:

* All adult, admitted patients of Covid-19/SARS-2 between March 2020 to September 2021 at Sultan Qaboos University Hospital

Exclusion Criteria:

* Patients with missing data or transferred to another hospital.
* The patients with chronic kidney disease and an estimated glomerular filtration rate (eGFR) of less than 30 mL/min/1.73m², or who underwent renal replacement therapy prior to admission

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to ICU with Covid-19 infection during the study period
Sampling Method: Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Acute Kidney Disease in Covid-19 patients admitted to ICU | up to 45 days
  Incidence of Acute Kidney Disease in Covid-19 patients admitted to ICU

SECONDARY OUTCOMES:
Association of glycemic status with Acute Kidney Injury in Covid-19 ICU cases. | Up to 45 days
  To study the association of glycemic status with Acute Kidney Injury in Covid-19 ICU cases.
Predictors and outcome of proportion of patients requiring renal replacement therapy | Up to 45 days
  To study the predictors and outcome of proportion of patients requiring renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Burad, MD, EDIC, Principal Investigator — Sultan Qaboos University Hospital
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after a few months of publication on Mendeley
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: IPD will be shared after a few months of Publication of the research
Access Criteria: Accessible to all
URL: https://data.mendeley.com

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Lowe R, Ferrari M, Nasim-Mohi M, Jackson A, Beecham R, Veighey K, Cusack R, Richardson D, Grocott M, Levett D, Dushianthan A; University Hospital Southampton Critical Care Team and the REACT COVID investigators. Clinical characteristics and outcome of critically ill COVID-19 patients with acute kidney injury: a single centre cohort study. BMC Nephrol. 2021 Mar 15;22(1):92. doi: 10.1186/s12882-021-02296-z. PMID 33722189
- [Background] Ghosn M, Attallah N, Badr M, Abdallah K, De Oliveira B, Nadeem A, Varghese Y, Munde D, Salam S, Abduljawad B, Saleh K, Elkambergy H, Wahla A, Taha A, Dibu J, Bayrlee A, Hamed F, Rahman N, Mallat J. Severe Acute Kidney Injury in Critically Ill Patients with COVID-19 Admitted to ICU: Incidence, Risk Factors, and Outcomes. J Clin Med. 2021 Mar 15;10(6):1217. doi: 10.3390/jcm10061217. PMID 33804100
- [Background] Pineiro GJ, Molina-Andujar A, Hermida E, Blasco M, Quintana LF, Rojas GM, Mercadal J, Castro P, Sandoval E, Andrea R, Fernandez J, Badia JR, Soriano A, Poch E; Hospital Clinic Critical Care COVID-19 working group (CCCC). Severe acute kidney injury in critically ill COVID-19 patients. J Nephrol. 2021 Apr;34(2):285-293. doi: 10.1007/s40620-020-00918-7. Epub 2021 Jan 2. PMID 33387345
- [Background] Khalili S, Sabaghian T, Sedaghat M, Soroureddin Z, Askari E, Khalili N. Prevalence, Risk Factors and Outcomes Associated with Acute Kidney Injury in Patients Hospitalized for COVID-19: A Comparative Study between Diabetic and Nondiabetic Patients. J Diabetes Res. 2021 Jan 6;2021:6666086. doi: 10.1155/2021/6666086. eCollection 2021. PMID 33506050
- [Background] Cau A, Cheng MP, Lee T, Levin A, Lee TC, Vinh DC, Lamontagne F, Singer J, Walley KR, Murthy S, Patrick D, Rewa O, Winston B, Marshall J, Boyd J, Russell JA. Acute Kidney Injury and Renal Replacement Therapy in COVID-19 Versus Other Respiratory Viruses: A Systematic Review and Meta-Analysis. Can J Kidney Health Dis. 2021 Oct 30;8:20543581211052185. doi: 10.1177/20543581211052185. eCollection 2021. PMID 34733538
- [Background] Nadim MK, Forni LG, Mehta RL, Connor MJ Jr, Liu KD, Ostermann M, Rimmele T, Zarbock A, Bell S, Bihorac A, Cantaluppi V, Hoste E, Husain-Syed F, Germain MJ, Goldstein SL, Gupta S, Joannidis M, Kashani K, Koyner JL, Legrand M, Lumlertgul N, Mohan S, Pannu N, Peng Z, Perez-Fernandez XL, Pickkers P, Prowle J, Reis T, Srisawat N, Tolwani A, Vijayan A, Villa G, Yang L, Ronco C, Kellum JA. COVID-19-associated acute kidney injury: consensus report of the 25th Acute Disease Quality Initiative (ADQI) Workgroup. Nat Rev Nephrol. 2020 Dec;16(12):747-764. doi: 10.1038/s41581-020-00356-5. Epub 2020 Oct 15. PMID 33060844
- [Background] Burke E, Haber E, Pike CW, Sonti R. Outcomes of renal replacement therapy in the critically ill with COVID-19. Med Intensiva (Engl Ed). 2021 Aug-Sep;45(6):325-331. doi: 10.1016/j.medine.2021.02.006. PMID 34294231